CLINICAL TRIAL: NCT07291154
Title: Impact of APP-assisted Patient Management on the Quality Control of Blood Purification Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunfeng Xia (Other)
Responsible Party: Sponsor-Investigator, Yunfeng Xia, Cheif physician, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1st ChongqingMedicalUniversity
Record Dates: First submitted 2025-09-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease (ESRD); Maintenance Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP management group (Experimental): For the APP management group, according to the specific conditions of patients such as age, gender, primary disease and complications, the "Yueya" mini-program and WeChat will be used to provide individualized and all-weather guidance for dialysis patients in their daily lives, including health knowledge education, diet and exercise guidance, medication supervision, condition monitoring and real-time feedback.
  Interventions: Behavioral: APP-based management
- Non-APP management group (No Intervention): For the non-APP management group, the APP mini-program will not be used to guide patients' daily lives, and only the previous routine management methods will be adopted.

INTERVENTIONS:
Behavioral: APP-based management — Based on patients' specific conditions such as age, gender, primary disease, and complications, the APP-based management will provide individualized and round-the-clock guidance for dialysis patients in their daily lives through the "Yueya" mini-program and WeChat. This guidance covers various aspects, including health knowledge education, diet and exercise guidance, medication supervision, condition monitoring, and real-time feedback.
  Arms: APP management group

SUMMARY:
Many maintenance hemodialysis (MHD) patients develop negative outlooks due to their illnesses and complications, making their quality of life and prognosis a clinical concern. Effective life management and treatment cooperation are crucial to improving dialysis quality and patient outcomes. This trial aims to evaluate whether management through the "Yueya" mini-program and WeChat can provide personalized guidance such as health education, diet, exercise, medication supervision, and condition monitoring to enhance treatment compliance, quality of life, strengthen quality control in the hemodialysis unit, and improve patient prognosis.

Patients will be divided into a group receiving support via the "Yueya" mini-program and WeChat, and a control group receiving routine care. Clinical and laboratory indicators, cardiovascular events, death, hospitalization, quality of life, and compliance will be recorded and compared between groups to assess the impact of APP-assisted patient management on the quality of MHD blood purification therapy and the prognosis of MHD patients.

DETAILED DESCRIPTION:
Affected by their own diseases and various complications, many maintenance hemodialysis (MHD) patients have a negative and pessimistic attitude toward life. Their quality of life and prognosis have always been a concern for clinicians. Therefore, how to adjust and manage the lives of these patients, enable them to actively cooperate with various treatment methods, maximize the quality of blood purification therapy, and improve their quality of life and prognosis has become an extremely important research topic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 5 chronic kidney disease, who have received maintenance hemodialysis for more than 3 months, are aged between 18 and 75 years old, and have regular dialysis three times a week.
* Patients with relatively stable condition, who are able to take care of themselves and willing to cooperate with the study.
* Patients who can understand and proficiently use WeChat and the "Yueya" mini - program used in this study.

Exclusion Criteria:

* Patients with communication barriers or other conditions that prevent them from cooperating with the study.
* Patients who have a history of acute myocardial infarction, cerebral infarction or intracerebral hemorrhage in the past six months.
* Patients who are not willing to actively cooperate with the study.
* Patients with severe liver cirrhosis, active tuberculosis and AIDS.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality rate | About 1 year
  In this study, mortality rate was used as a prognostic indicator.
Hospitalization rate | About 1 year
  In this study, the hospitalization rate was used as a prognostic indicator.
Kidney Disease Quality of Life | About 1 year
  Measuring the quality of life of hemodialysis patients through the Kidney Disease Quality of Life-36（KDQOL-36） scale. If the KDQOL-36 score increases, the quality of life is considered to be improved.
Incidence of cardiovascular events | About 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided